CLINICAL TRIAL: NCT03544047
Title: Clinical Study on Drug Sensitivity Verification or Prediction of Therapy for Breast Cancer by Patient-Derived Organoid Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Fei Ma, Professor, Peking Union Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC201804007
Record Dates: First submitted 2018-04-26; First posted 2018-06-01 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-05

CONDITIONS: Organoid
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Patient was first treated with paclitaxel (PTX) chemotherapy 3 cycles (2 weeks regimen) and Herceptin was treated in HER2 amplification patients. After 3 cycles. If the tumor continues to reduce in the first 3 cycles, continue paclitaxel chemotherapy for 3 cycles (6 weeks) and Herceptin was treated in HER2 amplification patients. If the evaluation of the curative effect is SD or PD, according to the result of drug sensitivity of the class organ, combined with the clinical practice, the doctor chooses the most sensitive treatment plan, and continues the 2 cycle treatment (6 weeks).
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Patient was first treated with paclitaxel (PTX) chemotherapy 3 cycles (2 weeks regimen). If the tumor continues to reduce in the first 3 cycles, continue paclitaxel chemotherapy for 3 cycles (6 weeks).

SUMMARY:
This is a single center, single arm, open and exploratory clinical study, with 50 cases planned for a period of 2 years. The purpose of this study is to evaluate the consistency and accuracy of Patient-Derived Organoid Model of breast cancer to predict the clinical efficacy of the drug, as well as the possibility of guiding the neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
After obtaining informed consent, patients who met the eligibility criteria underwent biopsy of the primary lesion or metastatic lesion (such as lymph node).Under the premise of ensuring normal detection requirements, a certain volume of fresh tumor tissues will be retained and used for the cultivation of Patient-Derived Organoid Model.If the organoid cultivation is not successful, the corresponding follow-up observation will be stopped.If the organoid cultivation is successful, drug sensitivity verification or prediction by Patient-Derived Organoid Model will be completed (final report will be available in about one month). During this period, the patient was first treated with paclitaxel (PTX) chemotherapy 3 cycles (2 weeks regimen) and Herceptin was treated in HER2 amplification patients. After 3 cycles, the efficacy was assessed according to the RECIST solid tumor evaluation standard (version 1.1), and the evaluation methods mainly included physical examination, ultrasound, CT and MRI.If the tumor continues to reduce in the first 3 cycles, continue paclitaxel chemotherapy for 3 cycles (6 weeks) and Herceptin was treated in HER2 amplification patients.If the evaluation of the curative effect is SD or PD, according to the result of drug sensitivity of the class organ, combined with the clinical practice, the doctor chooses the most sensitive treatment plan, and continues the 2 cycle treatment (6 weeks).After the completion of the evaluation, combined with the clinical situation, the next step is decided.For those who meet the conditions of the operation, the modified radical mastectomy or breast conserving surgery was performed after the neoadjuvant chemotherapy. The pCR status of the primary breast cancer and the axillary lymph nodes were evaluated after the operation. The adjuvant radiotherapy and endocrine therapy were given after the operation, and the long-term survival was observed.

Drug sensitivity tests include single drug and drug combination. The organs that are successfully cultured will be kept in liquid nitrogen for a specific time.

ELIGIBILITY:
Inclusion Criteria:

* The age is more than 18 years old;
* Pathology and immunohistochemical diagnosis of stage II-III breast cancer patients;
* No prior treatment (such as anti-tumor therapy, immunotherapy, related surgery, etc.) may affect the outcome of the treatment;
* According to the RECIST standard, the lesion was measured (the diameter of the primary lesion was greater than 1.0cm or the short diameter of the lymph node was greater than 1.5cm);
* Metastatic lesions or primary lesions can obtain surgical tissue or adequate biopsy tissue;
* No clinical diagnosis of other malignancies, unstable complications or uncontrolled infection;
* ECOG PS score: 0-2 points;
* Life expectancy is greater than 6 month;
* The main organ function is normal;
* The subjects volunteered to participate in this study, signed informed consent, followed up with good compliance.

Exclusion Criteria:

* Unable to obtain sufficient tumor organizer by operation or biopsy;
* Pregnant and lactating patients;
* Patients with peripheral nervous system disorder caused by disease or have significant mental disorders and history of central nervous system disorders;
* Patients with severe infections or active digestive tract ulcers need to be treated;
* Allergic to chemotherapy drugs or surgical contraindication;
* History of other malignant tumors;
* Severe liver disease (such as cirrhosis), cardiovascular disease, kidney disease, respiratory disease, blood system disease, or uncontrolled diabetes;
* Participating in or participating in other clinical trials within a month.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response rates (ORR) | up to 36 months
  Defined as complete response (CR) + partial response (PR), assessed based on Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria.

SECONDARY OUTCOMES:
Surgical excision rate | up to 36 months
  After neoadjuvant chemotherapy, the ratio of patients who achieved surgical resection.
Pathologic complete respons (pCR) rate | up to 36 months
  pCR is defined as no infiltrating tumor cells in pathological examination in the primary breast and axillary lymph nodes.
Disease-free survival (DFS) | up to 36 months
  The period after curative treatment when no disease can be detected)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided